CLINICAL TRIAL: NCT04407208
Title: Convalescent Plasma Therapy in Patients With COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biofarma (Industry)
Collaborators: Rumah Sakit Pusat Angkatan Darat Gatot Soebroto (Other); Eijkman Institute for Molecular Biology (Other)
Responsible Party: Principal Investigator, dr. Marliana Sri Rejeki, Sp.FK, Medical doctor, clinical pharmacologist, Biofarma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3471041S322342020040800002
Record Dates: First submitted 2020-05-16; First posted 2020-05-29 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Convalescence; Corona Virus Infection; Plaque
Keywords: COVID-19; convalescent plasma; treatment; severe ill
MeSH Terms: conditions — Convalescence; Coronavirus Infections; Plaque, Amyloid; COVID-19

STUDY DESIGN:
Intervention Model Description: single-arm, pre, and post-test dependent group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Convalescent plasma recipient (Experimental): Recipients receive 3 times of each 100 ml convalescent plasma on day 0, 3, and 6
  Interventions: Biological: Convalescent plasma

INTERVENTIONS:
Biological: Convalescent plasma — The minimum titer of specific antibody is 1/80

SUMMARY:
Scientists and medical workers all around the world were running out of time to manage COVID-19. Several studies have been done to understand the disease and ultimately to find possible treatment. Based on those studies, one of the potential treatment was antibody transfer from recovered COVID-19 patients. Passive antibody transfer was a fast and easy choice. The rational use of antibody from the patient's plasma is a natural neutralizing protein to the cell-infected virus and could possibly slow the active infection down. Investigators initiate an intervention study with purposes to produce quality convalescent plasma from the recovered patients, define the safety of plasma for human use and as an alternative treatment to improve the clinical outcomes of severe COVID-19 patients.

The study hypothesis is convalescent plasma is safe and could possibly improve outcome of severe (non-critical) COVID-19 patients. This research will conduct the plaque reduction neutralizing test (PRNT) of recipient blood in vitro. The plasma will be collected in the blood transfusion unit (BTU) in Gatot Soebroto hospital. The storage, testing, transfer, and transfusion of eligible convalescent plasma are the authority of Gatot Soebroto BTU. PRNT and plasma antibody titer measurement from donor plasma will be conducted at Eijkman Institute of Molecular Biology.

Investigators enroll approximately 10 patients consecutively, who will be admitted at Gatot Soebroto hospital. Baseline demographic characteristics of samples are recorded. Clinical dan laboratory data will be measured before and after plasma transfusion periodically. The measured variables are pharmacological therapy (antivirus, antibiotics, steroids), invasive oxygen therapy, oxygen index, sequential organ failure assessment (SOFA) score, and laboratory parameters such as leukocyte count, blood chemical panel include liver and renal function, C-reactive protein, procalcitonin, IL-6 and immunoglobulin titer of the recipient and also chest X-ray evaluation.

The potential expected risk of plasma transfusions is transfusion reaction (immunological or non-immune related) and transferred foreign pathogen. Investigator will report and treat all adverse events after plasma transfusion has been done. A severe adverse event (SAE) will also report in a special form to sponsor and data safety monitoring board (DSMB). There is theoretically antibody-dependent enhancement (ADE) mechanism from COVID-19 whom will receive plasma transfusion to progress to severe immune response.

This preliminary study is supposed to provide supporting data and experience of plasma processing to a larger study in the near future.

DETAILED DESCRIPTION:
The rational use of antibodies from the recovered patient's plasma as a natural neutralizing antibody to the cell-infected virus (plaques). Several expanded use of convalescent plasma therapy to severe and/or critically ill COVID-19 patients had been done in the US and China. Investigator reported that 5 patients received convalescent plasma, three patients were successfully discharged and 2 patients improved.

Based on the previous study, investigators initiate an intervention study with purposes to produce quality convalescent plasma from the recovered patients and to find an alternative treatment to improve the clinical outcomes of severe COVID-19 patients.

Investigators research questions are

1. Are the convalescent plasma could neutralize cell-infected virus in vitro?
2. Are those COVID-19 patients who received convalescent plasma will have a better prognosis and possibly be cured? The Investigator study hypothesis is convalescent plasma could possibly cure severe (non-critical) COVID-19 patients.

The primary objective of this study is to produce a good quality convalescent plasma from recovered COVID-19 patient which could neutralize the plaque in vitro and in Vivo. In Vivo neutralization will be monitored based on the patient's clinical improvement of symptoms, laboratory, and radiology assessment.

Invitro tests will be done to the recipient plasma before and after convalescent plasma transfusion. The objective evaluation will be a plaque reduction neutralizing test (PRNT) of recipient plasma. Donor plasma will be collected by apheresis methods at the Gatot Soebroto Blood transfusion unit (BTU).

All donors must meet the eligibility criteria and sign an informed consent form. Donor's plasma will be screened for blood-borne infection pathogens in BTU. Each donor will produce 210 ml of plasma, which 200 ml will be stored in 2 separate bags (each 100 ml) and 3 ml of plasma will be tested for antibody anti-COVID-19 titer in Biofarma and 3 ml of plasma will be tested for PRNT in Eijkman Institute. Plasma transfusion will be given to COVID-19 patients with severe (IIb) and critical conditions. The storage, testing, transfer, and transfusion of eligible convalescent plasma are the authority of Gatot Soebroto BTU. Investigators enroll approximately 10 patients consecutively, who will be admitted at Gatot Soebroto hospital.

All recipients will be enrolled consecutively if they met the eligibility criteria. Baseline demographic characteristics of the included patient are recorded in case report forms. Clinical and laboratory data will be measured before the plasma transfusion. Pre-transfusion patients will be put in group 1. Whereas group 2 is the same patient but received the convalescent plasma.

Transfusions will be given twice in 100 ml bag, during the 1st 4 hours, the acute adverse event will be monitored. There will be three serial transfusions, on the 1st day, 3rd day, and 6th day. The clinical, laboratory and radiology parameters will be re-measured after the14th day and they will be analyzed.

Data analysis will be done after all the measurement is finished and recorded in clinical report form. Investigators will find the mean difference of ordinal variables between group 1 and group two with the Wilcoxon signed-rank test (alternative to the paired T-test). The relative risk (risk reduction) of nominal variables will be measured between group 1 and group 2. Unfortunately, it is impossible to determine the number needed to harm (NNH) in this research since both groups are depending on each other.

All documents regarding the study will be kept in data form and will be protected with a password. We will concern about the safety of convalescent plasma by recording all adverse events after transfusion. To anticipate the risk of AE progression to a severe adverse event (SAE), all of the AE will be treated as soon as it is found according to the clinical competence of treating physicians. SAE will be reported in a certain form to sponsor and data safety monitoring board as soon as possible.

Investigators are all aware of the potential ethical issue regarding this study. The plasma convalescent is an alternative therapy for COVID-19, and urgently needed because of the pandemic situation currently happen. Investigators are weighing all potential expected and theoretical risks and benefits of convalescent plasma transfusion. The potential expected risk of plasma transfusions is transfusion reaction (immunological or non-immune related) and transferred unwanted pathogen. The theoretical risk from plasma transfusion of COVID-19 patient is an antibody-dependent enhancement (ADE) mechanism as seen in dengue patients. A Potential benefit of plasma for the patient is the neutralizing potential of a polyclonal antibody to cell infected SARS-Cov2. Resulting in faster recovery and improvement of the disease stages.

All donors will read the informed consent form thoroughly and willingly given their plasma draw at Gatot Soebroto BTU. The donor could revoke his/her consent at any time before being transfused, even after the plasma has been processed and stored in BTU. Donor's decision will not affect his/her future treatment at Gatot Soebroto hospital.

This preliminary study is supposed to provide supporting data and experience of plasma processing to a larger study in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 case with RT-PCR
* Stage IIb of COVID-19 or higher
* Consent was given by the patient or legal guardian

Exclusion Criteria:

* Pregnant
* History of anaphylactic reaction in previous blood product transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Plaque reduction neutralization test (PNRT) | day 7 after first transfusion
  PNRT50
D-dimer | day 1,4,7,14 after first transfusion
  Change of D-dimer compared between pre and post transfusion
C-Reactive Protein (CRP) | day 1,4,7,14 after first transfusion
  Change of CRP compared between pre and post transfusion
International Normalized Ratio (INR) | day 1,4,7,14 after first transfusion
  Change of INR compared between pre and post transfusion
Oxygenation Index | day 1,4,7,14 after first transfusion
  Change of OI compared between pre and post transfusion
Chest X-ray | day 1,4,7,28 after first transfusion
  Change of CXR with CXR covid score compared between pre and post transfusion

SECONDARY OUTCOMES:
severe adverse event | from day 0 to 14 days after plasma transfusion
  every adverse event that cause patient to die, prolonged hospitalization or worsening clinical stage of illness

CONTACTS AND LOCATIONS:
Overall Officials: Nana Sarnadi, Sp.OG, Study Director — director of research and develpment
Locations (1):
- Gatot Soebroto central army presidential hospital, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rejeki MS, Sarnadi N, Wihastuti R, Fazharyasti V, Samin WY, Yudhaputri FA, Johar E, Nurainy N, Bachtiar NS, Muljono DH. Convalescent plasma therapy in patients with moderate-to-severe COVID-19: A study from Indonesia for clinical research in low- and middle-income countries. EClinicalMedicine. 2021 Jun;36:100931. doi: 10.1016/j.eclinm.2021.100931. Epub 2021 Jun 4. PMID 34104878

DOCUMENTS (1):
  • Study Protocol (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT04407208/Prot_000.pdf